CLINICAL TRIAL: NCT05511051
Title: A Prospective Multi-centered Randomized Controlled Trial on Fruquintinib in Combination With Hepatic Arterial Infusion Chemotherapy (HAIC) in the Treatment of Liver Metastatic Colorectal Cancer After Failure of Second-line Systematic Therapy
Brief Title: A Prospective Multi-centered Randomized Controlled Trial on Fruquintinib in Combination With HAIC in the Treatment of Liver Metastatic Colorectal Cancer After Failure of Second-line Systematic Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Principal Investigator, Yue Han, Chief physician, Interventional Therapy Department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-N1-CRC102
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: Third-line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib + HAIC (Experimental): Fruquintinib: 5 mg orally once daily for 21 days on followed by 7 days off (q4w); HAIC: oxaliplatin 100 mg/m2, leucovorin calcium 200 mg/m2, fluorouracil 2000 mg/m2 24-hour drip, q4w, 2 cycles; HAIC treatment was administered during fruquintinib rest; HAIC was discontinued 1 day before surgery, on the day of completion of surgery, and 5 days after surgery;
  Interventions: Drug: Fruquintinib; Drug: HAIC
- Fruquintinib (Active Comparator): Fruquintinib: 5 mg orally once daily for 21 days on followed by 7 days off (q4w);
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib
Drug: HAIC — HAIC
  Arms: Fruquintinib + HAIC

SUMMARY:
The current study is to investigate the safety and efficacy of fruquintinib combined with HAIC in patients with advanced colorectal liver metastases who have failed second-line systemic standard treatment, in order to provide more survival opportunities for the second progression of advanced colorectal liver metastases.

DETAILED DESCRIPTION:
Among Chinese colorectal cancer patients, 43.8% had metastasis at the time of diagnosis, of which liver metastasis accounted for 51.5%. In addition, it was reported that 10%-25% of patients developed liver metastasis after radical resection of colorectal cancer, and more than two-thirds of colorectal patients eventually developed liver metastasis. Colorectal liver metastasis was reported to be the most important cause of death in colorectal cancer patients.The median survival time of untreated liver metastases was only 6.9 months, and the 5-year survival rate of unresectable patients was less than 5%, and for unresectable colorectal liver metastasis, the median survival time could reach 30.9 months after comprehensive treatment.

Fruquintinib, a VEGFR 1/2/3 inhibitor, is one of the standard 3rd-line therapy for colorectal cancer, which has already been approved and marketed in China. In phase III FRESCO study, liver metastases subgroup showed that the median OS of fruquintinib group was 8.61 months, which was 2.63 months longer than that of control group, reducing death risk by 41%, with statistically significant P value.

Patients with large tumor burden mainly caused by liver metastasis and with insignificant or refractory response to drug therapy, or patients who cannot tolerate systemic therapy, can be combined with transcatheter arterial chemoembolization (HAI) or transcatheter arterial chemoembolization (TACE) at appropriate time, which helps to prolong the progression-free time and overall survival.

The current study is to investigate the safety and efficacy of fruquintinib combined with HAIC in patients with advanced colorectal liver metastases who have failed second-line systemic standard treatment, in order to provide more survival opportunities for the second progression of advanced colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Age ≥ 18 years;
3. Patients with unresectable colorectal liver metastases who have failed standard second-line systemic therapy, who have not previously received HAIC therapy, and have not received third-line standard targeted agents (regorafenib or fruquintinib or trifluridine tipiracil (TAS-102);
4. Definition of liver metastases: at least 1 measurable liver metastasis lesion (based on RECIST 1.1); if the liver metastases are single, the tumor is > 5 cm; if multiple tumors, it needs to be greater than or equal to 4, of which at least 1 exceeds 3 cm;
5. PFS > 4 months from last dose of oxaliplatin with FOLFOX regimen
6. Child-Pugh classification of liver function: A;
7. ECOG performance status 0-1, and no deterioration within 7 days;
8. BMI ≥ 18;
9. Expected survival ≥ 3 months;
10. Vital organs function in accordance with the following requirements (any blood components and cell growth factors are not allowed within 14 days before enrollment):

    * Absolute neutrophil count ≥ 1.5 × 109/L and white blood cells ≥ 4.0 × 109/L;
    * Platelets ≥ 100 × 109/L;
    * Hemoglobin ≥ 90 g/L;
    * Total bilirubin TBIL ≤ 1.5 times ULN;
    * ALT and AST ≤ 5 times ULN;
    * Urea nitrogen/urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN (and creatinine clearance (CCr) ≥ 50 mL/min);
    * Left ventricular ejection fraction (LVEF) ≥ 50%;
    * Fridericia-corrected QT interval (QTcF) < 470 milliseconds.
    * INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
11. women of childbearing age need to take effective contraceptive measures;
12. good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Unable to comply with the study protocol or study procedures;
2. Pregnant or breastfeeding women;
3. Any factor affecting oral administration;
4. Evidence of central nervous system metastases;
5. Concurrent with any of the following: uncontrolled hypertension, coronary artery disease, arrhythmia, and heart failure;
6. Alcohol or drug abuse within 4 weeks after the last clinical trial;
7. Previous VEGFR inhibition therapy;
8. Uncontrolled severe concurrent infection resulting in disability;
9. Proteinuria ≥ 2 + (1.0 g/24 h);
10. Evidence or history of bleeding tendency within 2 months prior to enrollment, regardless of seriousness;
11. Arterial/venous thromboembolic events, such as cerebrovascular accidents (including transient ischemic attack), within 12 months before the first treatment;
12. Acute myocardial infarction, acute coronary syndrome or CABG within 6 months before the first treatment;
13. Fractures or wounds that have not been cured for a long time;
14. coagulopathy, bleeding tendency or receiving anticoagulant therapy;
15. Inactivated vaccines within 4 weeks prior to enrollment or possible during the study;
16. Patients with other malignant tumors within 5 years before enrollment, except for basal cell or squamous cell carcinoma of the skin after radical resection, or cervical carcinoma in situ;
17. Active autoimmune diseases or history of autoimmune diseases within 4 weeks before enrollment;
18. Previous allogeneic bone marrow transplantation or organ transplantation;
19. Subjects who are allergic to the study drug or any of its adjuvant preparations;
20. Electrolyte abnormalities judged clinically significant by the investigator;
21. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must have excluded active HBV infection, ie, positive HBV DNA (> 1 × 104 copies/mL or > 2000 IU/mL); known hepatitis C virus (HCV) infection and positive HCV RNA (> 1 × 103 copies/mL);
22. Unresolved toxicities above CTCAE v5.0 grade 1 due to any prior anticancer therapy, excluding alopecia, lymphopenia, and oxaliplatin-induced neurotoxicity ≤ grade 2;
23. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 28 days before enrollment;
24. with brain metastases, or with severe malignant pleural effusion and ascites;
25. Any other diseases, clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the investigator 's judgment, there is reason to suspect that the patient has a disease or condition that is not suitable for the use of the study drug (such as having seizures and requiring treatment), or will affect the interpretation of the study results, or put the patient at high risk;
26. Patients who are considered unsuitable for inclusion in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from randomization until death due to any cause, assessed up to 2 year
  every two months after end of treatment (EOT) observation period at 30 days after the last medication every two months after end of treatment (EOT) observation period at 30 days after the last medication every two months after end of treatment (EOT) observation period at 30 days after the last medication

SECONDARY OUTCOMES:
Progress-free Survival | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Objective Response Rate | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to within 30 days after the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Dalian Medial University Affiliated Second Hospital, Dalian
  - People's Hospital of Inner Mongolia, Hohhot

IPD SHARING:
Plan to Share IPD: No